CLINICAL TRIAL: NCT05986773
Title: Diuretic Strategies in Acute Heart Failure Patients at High Risk for Diuretic Resistance (P-Value-AHF): A Multicentre, Randomized, Parallel-group, Open-label Trial
Brief Title: Diuretic Strategies in Acute Heart Failure Patients at High Risk for Diuretic Resistance
Acronym: P-Value-AHF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment in both centers
Sponsor: Stadtspital Zürich (Other)
Collaborators: Ospedale Regionale di Lugano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Value-AHF
Record Dates: First submitted 2023-04-27; First posted 2023-08-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Acute Heart Failure; Diuretic Resistance
Keywords: Diuretic therapy
MeSH Terms: interventions — Furosemide; Metolazone; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group FF (Active Comparator): Group FF will receive a doubled dose Furosemide i.v.
  The first standard dose Furosemide i.v. should be administered according to the current guidelines: (i) diuretic-naïve patients should receive Furosemide 40 mg i.v.; (ii) patients on a maintenance oral diuretic treatment should receive the equivalent dose i.v.
  Study medications will be used according to the prescribing information: Furosemide will be administered as an intravenous injection.
  Interventions: Drug: Furosemide
- group FM (Active Comparator): Group FM will receive a combination of standard dose Furosemide i.v. and Metolazone 5 mg p.o.
  The first standard dose Furosemide i.v. should be administered according to the current guidelines: (i) diuretic-naïve patients should receive Furosemide 40 mg i.v.; (ii) patients on a maintenance oral diuretic treatment should receive the equivalent dose i.v.
  Study medications will be used according to the prescribing information: Furosemide will be administered as an intravenous injection. Metolazone will be administered orally.
  Interventions: Drug: Furosemide; Drug: Metolazone
- group FA (Active Comparator): Group FA will receive a combination of standard dose Furosemide i.v. and Acetazolamide 500 mg i.v.
  The first standard dose Furosemide i.v. should be administered according to the current guidelines: (i) diuretic-naïve patients should receive Furosemide 40 mg i.v.; (ii) patients on a maintenance oral diuretic treatment should receive the equivalent dose i.v.
  Study medications will be used according to the prescribing information: Furosemide will be administered as an intravenous injection. Acetazolamide (500mg) will be administered intravenously as a short infusion.
  Interventions: Drug: Furosemide; Drug: Acetazolamide

INTERVENTIONS:
Drug: Furosemide — Two to five hours after the initial standard dose Furosemide i.v, the patients are randomized towards 3 study-specific diuretic regimens: the first group will receive a doubled dose Furosemide i.v. (group FF), the second group will receive a combination of standard dose Furosemide i.v. and Metolazone 5 mg p.o. (group FM), the third group will receive a combination of standard dose Furosemide i.v. and Acetazolamide 500 mg i.v. (group FA).
  Other Names: Furosemide, doubled dose
Drug: Metolazone — Two to five hours after the initial standard dose Furosemide i.v, the patients are randomized towards 3 study-specific diuretic regimens: the first group will receive a doubled dose Furosemide i.v. (group FF), the second group will receive a combination of standard dose Furosemide i.v. and Metolazone 5 mg p.o. (group FM), the third group will receive a combination of standard dose Furosemide i.v. and Acetazolamide 500 mg i.v. (group FA).
  Other Names: Furosemide + Metolazone
  Arms: group FM
Drug: Acetazolamide — Two to five hours after the initial standard dose Furosemide i.v, the patients are randomized towards 3 study-specific diuretic regimens: the first group will receive a doubled dose Furosemide i.v. (group FF), the second group will receive a combination of standard dose Furosemide i.v. and Metolazone 5 mg p.o. (group FM), the third group will receive a combination of standard dose Furosemide i.v. and Acetazolamide 500 mg i.v. (group FA).
  Other Names: Furosemide + Acetazolamide
  Arms: group FA

SUMMARY:
The P-VALUE-AHF trial is a multicenter, randomized, open-label, parallel-group trial on the diuretic and decongestive effects of different diuretic escalation strategies in patients with acute heart failure and diuretic resistance.

The main aims are

* to compare the diuretic efficacy of three therapeutic strategies in patients with acute heart failure and diuretic resistance.
* to assess the improvement in clinical congestion and to compare the symptom-relief among the different treatment regimens

DETAILED DESCRIPTION:
The P-VALUE-AHF trial is a multicenter, randomized, open-label, parallel-group trial on the diuretic and decongestive effects of different diuretic escalation strategies in patients with acute heart failure (AHF) and diuretic resistance (DR).

Consenting patients with AHF and DR will be will be randomized towards 3 diuretic regimens. Two to five hours after the initial standard dose Furosemide i.v,

* the first group will receive a doubled dose Furosemide (group FF)
* the second group will receive a combination of standard dose Furosemide and Metolazone (group FM)
* the third group will receive a combination of standard dose Furosemide and Acetazolamide (group FA)

Objectives

* The primary objective is to compare the diuretic efficacy (measured as natriuresis and urine volume) of three therapeutic strategies in patients with acute heart failure and diuretic resistance.
* The secondary objective is to assess the improvement in clinical congestion (EVEREST congestion score) and to compare the symptom-relief (improvement of dyspnoea (VAS)) among the different treatment regimens (FF vs. FM vs. FA).

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergency hospital admission with clinical diagnosis of acute heart failure
* One or more clinical signs of volume overload (i.e., peripheral edema, pleural effusion, jugular venous distension)
* Low diuretic efficacy in the first 2 hours after the standard screening dose Furosemide i.v. (i.e., urine volume < 300 ml and urine sodium concentration < 70 mmol/L)
* Plasma N terminal-proBNP level at enrolment > 1000 ng/L
* Signed Informed Consent form

Exclusion Criteria:

* Maintenance treatment with Acetazolamide or Metolazone
* Use of any non-protocol defined diuretic agent that cannot be stopped upon study inclusion except for sodium-glucose co-transporter-2 inhibitors (e.g., dapagliflozin, empagliflozin, canagliflozin) and mineralocorticoid receptor antagonists (e.g., spironolactone, eplerenone)
* Systolic blood pressure < 90 mmHg
* Expected use of intravenous vasopressors (e.g., noradrenaline, adrenaline), inotropes (e.g., dobutamine, milrinone, levosimendan) at any time point during the study
* Severe chronic kidney disease (estimated glomerular filtration rate < 15 ml/min/1.73 m2) or use of renal replacement therapy at any time before study inclusion
* Severe liver dysfunction or cirrhosis at risk of hepatic encephalopathy
* Severe electrolyte disturbances or metabolic acidosis requiring specific intravenous treatment
* Concurrent diagnosis of acute coronary syndrome requiring urgent revascularization
* History of cardiac transplantation or ventricular assist device
* Allergy, intolerance or other contraindication against one of the study drugs
* Pregnancy or breastfeeding
* Age below 18 years.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Diuretic efficacy after 6h | 6 hours after administration of the study-specific diuretic regimen
  urine- natrium concentration (mmol/L)

SECONDARY OUTCOMES:
Diuretic efficacy after 2h | 2 hours after administration of the study-specific diuretic regimen
  urine- natrium concentration (mmol/L)
Diuretic efficacy after 24h | 24 hours after administration of the study-specific diuretic regimen
  urine- natrium concentration (mmol/L)
Change in clinical congestion | 0 and 24 hours after administration of the study-specific diuretic regimen
  EVEREST congestion score
Change in dyspnea severity | 0 and 24 hours after administration of the study-specific diuretic regimen.
  numeric rating scale

OTHER OUTCOMES:
Safety Outcomes 1 | 0-24 hours after administration of the study-specific diuretic regimen
  Hypotension (SBP< 90 mmHg) with symptoms or requiring therapeutic intervention
Safety Outcomes 2 | 0-24 hours after administration of the study-specific diuretic regimen
  Increase in serum creatinine >50% from baseline
Safety Outcomes 3 | 0-24 hours after administration of the study-specific diuretic regimen
  New electrolyte disturbances (sodium < 130mmol/l or > 150mmol/l, potassium < 3.0mmol/l or > 5.5 mmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Arrigo, PD, Dr. med., Principal Investigator — City Hospital Zürich Triemli, Birmensdorferstr. 497, 8063 Zürich, Switzerland
Locations (1):
- Stadtspital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No